CLINICAL TRIAL: NCT00016874
Title: A Phase I Study Of 3-Aminopyridine-2-Carboxaldehyde Thiosemicarbazone (3-AP, Triapine) In Combination With Cisplatin And Paclitaxel In Patients With Advanced And Metastatic Cancer
Brief Title: 3-AP Plus Cisplatin and Paclitaxel in Treating Patients With Advanced or Metastatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vion Pharmaceuticals (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: VION-CLI-015; CDR0000068591 (Registry Identifier: PDQ (Physician Data Query)); AECM-1200012380; NCI-V01-1658
Record Dates: First submitted 2001-06-06; First posted 2003-09-09 (Estimated); Last update posted 2013-07-18 (Estimated); Status verified 2007-12

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Cisplatin; Paclitaxel; 3-aminopyridine-2-carboxaldehyde thiosemicarbazone

INTERVENTIONS:
Drug: cisplatin
Drug: paclitaxel
Drug: triapine

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of combining 3-AP, cisplatin, and paclitaxel in treating patients who have advanced or metastatic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the safety and tolerability of 3-AP, cisplatin, and paclitaxel in patients with advanced or metastatic cancer.
* Determine the toxic effects of this regimen in these patients.
* Determine the maximum tolerated dose and recommended phase II dose of this regimen in these patients.
* Determine the pharmacokinetic parameters of this regimen in these patients.
* Determine the tumor response in patients treated with this regimen.

OUTLINE: This is a dose-escalation study.

Patients receive 3-AP IV continuously over 96 hours on days 1-4 and paclitaxel IV over 3 hours followed by cisplatin IV over 1 hour on day 3. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients achieving complete response (CR) receive 1 additional course of therapy after documented CR. Patients with partial response or stable disease may receive therapy for up to 6 months.

Cohorts of 1-6 patients receive escalating doses of 3-AP, paclitaxel, and cisplatin until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity.

PROJECTED ACCRUAL: Approximately 25-30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed progressive advanced or metastatic cancer

  * Failed 1 or more prior standard therapies for disease OR
  * Unlikely to respond to any currently available therapies
* Measurable or evaluable disease
* No active CNS metastases

  * Previously treated CNS metastases allowed if no evidence of new CNS metastases and stable for at least 2 months

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-1

Life expectancy:

* More than 3 months

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 10 g/dL (transfusion allowed)
* No active bleeding or coagulation disorder (occult blood for gastrointestinal cancer allowed)

Hepatic:

* Bilirubin no greater than 1.5 mg/dL
* ALT/AST no greater than 3 times upper limit of normal (ULN) (5 times ULN if liver metastases present)
* Alkaline phosphatase no greater than 3 times ULN (5 times ULN if liver metastases present)
* Albumin at least 3.0 g/dL
* PT/PTT no greater than 1.5 times ULN

Renal:

* Creatinine no greater than 1.5 mg/dL

Cardiovascular:

* No active heart disease
* No myocardial infarction within the past 3 months
* No symptomatic coronary artery disease, heart block, or uncontrolled congestive heart failure

Pulmonary:

* No moderate to severe compromise in pulmonary function

Other:

* No mental deficits and/or psychiatric history that would preclude study
* No active infection
* No pre-existing severe hearing impairment
* No pre-existing grade 2 or greater neuropathy
* No prior severe allergic reaction to study drugs
* No other life-threatening illness
* No chronic toxic effects from prior chemotherapy greater than grade I
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 18 months after study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Concurrent hematopoietic growth factors allowed except if used prophylactically during first course of study therapy

Chemotherapy:

* More than 3 weeks since prior chemotherapy (6 weeks for nitrosourea or mitomycin) and recovered
* More than 6 months since prior combination cisplatin and paclitaxel
* Prior cisplatin or paclitaxel as single agents allowed
* Prior 3-AP allowed

Endocrine therapy:

* Not specified

Radiotherapy:

* More than 3 weeks since prior radiotherapy and recovered
* Concurrent radiotherapy to a single site of progressive disease allowed if site requires treatment within the first course of study therapy

Surgery:

* Not specified

Other:

* More than 3 weeks since any therapy for malignancy and recovered
* No other concurrent investigational drugs without consent of sponsor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-12; Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mario Sznol, MD, Study Chair — Vion Pharmaceuticals
Locations (2):
- United States (2):
  - New York Presbyterian Hospital - Cornell Campus, New York, New York
  - Albert Einstein Comprehensive Cancer Center, The Bronx, New York